CLINICAL TRIAL: NCT05400538
Title: Probiotics as Adjunct to Non Surgical Periodontal Therapy for Pregnant Women Domiciliary Oral Hygiene.
Brief Title: Probiotics as Adjunct to Non Surgical Periodontal Therapy for Pregnant Women Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-PREGNANCY
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Periodontal Diseases
Keywords: pregnancy
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial group (Experimental): Biorepair Toothpaste + Mousse domiciliary use
  Interventions: Other: Biorepair Toothpaste + Mousse
- Control group (Active Comparator): Biorepair Toothpaste domiciliary use.
  Interventions: Other: Biorepair Toothpaste

INTERVENTIONS:
Other: Biorepair Toothpaste + Mousse — Domiciliary application of the products twice a day.
  Arms: Trial group
Other: Biorepair Toothpaste — Domiciliary application of the product twice a day.
  Arms: Control group

SUMMARY:
The aim of the present study is to evaluate the use of probiotics in domiciliary oral hygiene procedures in pregnant women.

Patients consenting to participate to the study will undergo periodontal evaluation at the baseline (T0). Then, professional dental hygiene will be performed. Patients will be randomly assigned to:

* Trial group: home oral application of Biorepair Peribioma Toothpaste + Biorepair Peribioma mousse twice a day
* Control group: home oral application of Biorepair Peribioma Toothpaste

Patients will be evaluated after 1 month (T1), 3 (T2) and 6 (T3) months.

DETAILED DESCRIPTION:
The aim of the present study is to evaluate the use of probiotics in domiciliary oral hygiene procedures in pregnant women.

Patients consenting to participate to the study will undergo periodontal evaluation at the baseline (T0). Then, professional dental hygiene will be performed. Patients will be randomly assigned to:

* Trial group: home oral application of Biorepair Peribioma Toothpaste + Biorepair Peribioma mousse twice a day
* Control group: home oral application of Biorepair Peribioma Toothpaste

Patients will be evaluated after 1 month (T1), 3 (T2) and 6 (T3) months, the following indexes will be assessed: Probing Pocket Depth, Bleeding on Probing (percentage), Clinical Attachment Loss, Gingival recession, Plaque Control Record, Modified Gingival Index, Papillary Marginal Gingival Index.

ELIGIBILITY:
Inclusion Criteria:

* women at the 4th month of pregnancy

Exclusion Criteria:

* presence of cardiac pacemaker
* neurological and psychiatric diseases
* patients taking bisphosphonates during the previous 12 months from the beginning of the study
* patients undergoing anticancer therapy.
* patients with poor compliance.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Change in PPD - Probing Pocket Depth | Baseline, after 1, 3 and 6 months.
  Evaluation (in mm) of the depth of the gingival sulcus, through a millimeter periodontal probe; it is detected from the gingival margin to the bottom of the gingival sulcus or periodontal pocket, evaluated at 6 sites.
Change in BOP - Bleeding on Probing (percentage) | Baseline, after 1, 3 and 6 months.
  Site-specific assessment of the presence or absence of gum bleeding after the insertion of the periodontal probe for the detection of PPD, detected on 6 sites.
  Percentage of sites with bleeding on probing determines the BOP%.
Change in CAL - Clinical Attachment Loss | Baseline, after 1, 3 and 6 months.
  Measurement (in mm) of the position of the gingival margin in relation to the cemento-enamel junction (CEJ).
Change in R - Gingival recession | Baseline, after 1, 3 and 6 months.
  Distance (in mm) between the gingival margin and the amelo-cemental junction.
Change in PCR% - Plaque Control Record | Baseline, after 1, 3 and 6 months.
  % assessment of the amount of plaque on dental surfaces; it is detected on 4 surfaces: distal, mesial, vestibular, lingual / palatal. The number of sites with plaque is divided by the total number of sites available in the mouth and multiplied by 100. Results indicate the index as a percentage.
Change in MGI - Modified Gingival Index | Baseline, after 1, 3 and 6 months.
  Scoring criteria:
  * 0: normal
  * 1: mild inflammation (slight changes in color and texture, but not in all portions of gingival marginal or papillary)
  * 2: mild inflammation (slight changes in color and texture in all portions of gingival marginal or papillary)
  * 3: moderate (bright surface inflammation, erythema, edema, and/or hypertrophy of gingival marginal or papillary)
  * 4: severe inflammation (erythema, edema, and/or marginal gingival hypertrophy of the unit or spontaneous bleeding, papillary, congestion, or ulceration)
Change in PMGI - Papillary Marginal Gingival Index | Baseline, after 1, 3 and 6 months.
  Numerical score from 0 to 3 of gingival inflammation. Papille and gingival margins (vestibular and lingual) are given a score from 0 to 3. The score is given by the total amount of inflamed sites on the total of examined sites.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, MS, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.